CLINICAL TRIAL: NCT05463900
Title: Microbial and Human Determinants of the Onset of IBD Flares on a National Scale - an Observational Study
Brief Title: Microbial and Human Determinants of the Onset of IBD Flares
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Viome (Industry)
Responsible Party: Sponsor
Other Study IDs: V304
Record Dates: First submitted 2022-07-05; First posted 2022-07-19 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Ulcerative Colitis; Crohn Disease; Irritable Bowel; Crohns Disease Aggravated; Crohn Disease in Remission
Keywords: IBD; flare; UC; CD; HBI; SCCAI; stool; diarrhea; abdominal pain; inflammation; colon; rectum
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Irritable Bowel Syndrome; Diarrhea; Abdominal Pain; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ulcerative Colitis (UC): Individuals with an ICD-10 diagnosis of Ulcerative Colitis.
- Crohn's Disease (CD): Individuals with an ICD-10 diagnosis of Crohn's Disease.

SUMMARY:
This is a longitudinal, observational study that aims to identify the microbial and human molecular triggers of IBD flares via stool, saliva, and blood metatranscriptomes, whole blood proteome, and collected clinical metadata. This study is direct to participant and will not utilize clinical sites.

DETAILED DESCRIPTION:
This is a longitudinal, observational study that aims to identify the microbial and human molecular triggers of IBD flares via stool, saliva, and blood metatranscriptomes, whole blood proteome, and collected clinical metadata. This study will last approximately 3 years and will recruit up to 1000 Crohn's Disease participants and up to 1000 Ulcerative Colitis participants that will participant in the study for approximately 12 months. Participants will be sent at home sample collection kits and a study survey each month. If the survey responses indicate a participant is in a flare, they will be sent a sample collection kit and survey on a weekly basis until the flare is over and the monthly schedule resumes. The objective of the data analysis is to identify microbial functions that are predictive of the onset of a flare.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to provide written informed consent prior to screening
* Established diagnosis of small bowel or colonic Crohn's Disease (CD) or Ulcerative Colitis (UC)

Exclusion Criteria:

* Pregnant or breastfeeding
* Use of antibiotics within the last 3 months
* Bowel surgery in the past 3 months or planned bowel surgery during the 12-month study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of up to 1000 Ulcerative Colitis participants and up to 1000 Crohn's Disease participants that are 18 years of age or older and that meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Names of species | 3 years
  Species present in samples taken in IBD and IBD flare onset states.
Number of species | 3 years
  Number of each species present in sample taken in IBD and IBD flare onset states.

CONTACTS AND LOCATIONS:
Overall Officials: Momchilo Vuyisich, Principal Investigator — Viome
Locations (1):
- Viome Life Sciences, Bothell, Washington, United States